CLINICAL TRIAL: NCT04593888
Title: Gluten Reduction After Infancy and Risk of Celiac Disease
Brief Title: Gluten Reduction and Risk of Celiac Disease
Acronym: GRAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-00446
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Celiac Disease in Children; Autoimmune Diseases; type1diabetes
Keywords: gluten; diet
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Masking Description: study participants will be randomized to either the "gluten-reduced" or "no intervention" arm on-going after enrolment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): The group will be followed without any intervention, with regular visits at the research clinic.
- Gluten reduced diet (Experimental): Subjects will follow a diet that does not exceed a daily intake of 3 gram gluten.
  The group will be followed with regular visits at the research clinic.
  Interventions: Behavioral: Gluten reduced diet

INTERVENTIONS:
Behavioral: Gluten reduced diet — Dietary advice focusing on reducing gluten intake in children
  Arms: Gluten reduced diet

SUMMARY:
Celiac disease shares many features of other autoimmune diseases such as type 1 diabetes. Recently, it was published that higher amounts of gluten intake increased the risk for celiac disease. Optimal amounts of gluten to be introduced during weaning have not yet been established. The aim is to investigate if a gluten-restricted diet (e.g. below 3 gram per day) during the first 3 years of life will reduce the risk of develop CDA and IA in genetically predisposed children by the age of 7 years. Children who screened positive for HLA DQ2/X (X is neither DQ2 nor DQ8) in the GPPAD-02 (ASTR1D [ClinicalTrials.gov Identifier NCT03316261]) screening will be contacted by a study nurse.

DETAILED DESCRIPTION:
Gluten is a complex mixture of proteins, mainly gliadin and glutenin, rich in proline and glutamine amino acids which make these proteins resistant to complete degradation by enzymes in the small intestinal. Intolerance to gluten leads to inflammation of the intestinal epithelium and villous atrophy, a disorder called celiac disease. Celiac disease shares many features of other autoimmune diseases such as type 1 diabetes (T1D). First, celiac disease is associated with certain HLA genotypes of whom 95% of all patients with celiac disease carry the haplotypes DQA1*0501-DQB1*0201 (abbreviated DQ2) and the reminder 5% DQA1*0301-DQB1*0302 (abbreviated DQ8). There is a gene dose effect of HLA-DQ on the risk of develop celiac disease; 20% of the children homozygous for HLA-DQ2/DQ2 will develop celiac disease by 10 years of age. Second, celiac disease is also strongly associated with the presence of autoantibodies directed against tissue transglutaminase (tTGA) that occurs in 100% of children with celiac disease. Timing of gluten introduction and breastfeeding duration have previously been proposed to influence risk for celiac disease. However, based on the results from the multinational birth cohort study The Environmental determinants of Diabetes in the Young (TEDDY) study and other observational studies, timing of gluten introduction seems not associated with celiac disease in genetically at-risk children. In an RCT, introduction of small amounts of gluten at the age of 4-6 months did not reduce the risk for celiac disease by the age of 3 years in genetically at-risk children. Current international infant feeding recommendations recommend that gluten is introduced into the infant's diet anytime between 4-12 months of age and that consumption of large quantities of gluten should be avoided during the first month after gluten introduction and during infancy. Recently, the TEDDY study published that higher amounts of gluten intake increased the risk for celiac disease, which have been confirmed in two other observational cohort studies. In the TEDDY study, daily gluten intake was associated with higher increased risk of developing persistently positive tTGA, a definition coined celiac disease autoimmunity (CDA), as well as with celiac disease for every 1-g/day increase in gluten intake. Optimal amounts of gluten to be introduced during weaning have not yet been established. It is well known that an overlap between celiac disease and T1D exists most likely due to shared genetic risks of HLA-DQ2 and/or DQ8 in both disorders. Prospective studies in infants genetically predisposed to T1D and celiac disease showed that antibody positivity to both disorders begins in the first 1-3 years of life. The study aim is to investigate if a gluten-restricted diet during the first 3 years of life will reduce the risk of develop CDA and IA in genetically predisposed children by the age of 7 years.

ELIGIBILITY:
Inclusion Criteria:

* children screened positive for HLA DQ2/X (X is neither DQ2 or DQ8)
* children who refused enrolment to the on-going study PreSiCe (ClinicalTrials.gov Identifier NCT03562221)

Exclusion Criteria:

* congenital chronic disorder where intervention with diet may be affected
* written informed consent from both caregivers are missing

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1141 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Celiac disease autoimmunity (CDA) | from 6 months of age up until 7 years of age
  Children tested positive for tissue transglutaminase autoantibodies (tTGA) in two consecutive serum samples 3-6 months apart.

SECONDARY OUTCOMES:
Celiac disease (CD) | from 6 months of age up until 7 years of age
  celiac disease diagnosed, defined by intestinal biopsy showing a Marsh score of >2 or by high levels of tTGA with symptoms.

OTHER OUTCOMES:
Islet autoimmunity | from 6 months of age up until 7 years of age
  Children tested positive for typ1 1 diabetes related autoantibodies (IAA, GADA, IA2A) in two consecutive serum samples 3-6 months apart.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Agardh, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Clinical Research Center (CRC), Bldng 60:11, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andren Aronsson C, Lee HS, Hard Af Segerstad EM, Uusitalo U, Yang J, Koletzko S, Liu E, Kurppa K, Bingley PJ, Toppari J, Ziegler AG, She JX, Hagopian WA, Rewers M, Akolkar B, Krischer JP, Virtanen SM, Norris JM, Agardh D; TEDDY Study Group. Association of Gluten Intake During the First 5 Years of Life With Incidence of Celiac Disease Autoimmunity and Celiac Disease Among Children at Increased Risk. JAMA. 2019 Aug 13;322(6):514-523. doi: 10.1001/jama.2019.10329. PMID 31408136
- [Result] Marild K, Dong F, Lund-Blix NA, Seifert J, Baron AE, Waugh KC, Taki I, Stordal K, Tapia G, Stene LC, Johnson RK, Liu E, Rewers MJ, Norris JM. Gluten Intake and Risk of Celiac Disease: Long-Term Follow-up of an At-Risk Birth Cohort. Am J Gastroenterol. 2019 Aug;114(8):1307-1314. doi: 10.14309/ajg.0000000000000255. PMID 31082869
- [Result] Vriezinga SL, Auricchio R, Bravi E, Castillejo G, Chmielewska A, Crespo Escobar P, Kolacek S, Koletzko S, Korponay-Szabo IR, Mummert E, Polanco I, Putter H, Ribes-Koninckx C, Shamir R, Szajewska H, Werkstetter K, Greco L, Gyimesi J, Hartman C, Hogen Esch C, Hopman E, Ivarsson A, Koltai T, Koning F, Martinez-Ojinaga E, te Marvelde C, Pavic A, Romanos J, Stoopman E, Villanacci V, Wijmenga C, Troncone R, Mearin ML. Randomized feeding intervention in infants at high risk for celiac disease. N Engl J Med. 2014 Oct 2;371(14):1304-15. doi: 10.1056/NEJMoa1404172. PMID 25271603
- [Result] Lionetti E, Castellaneta S, Francavilla R, Pulvirenti A, Tonutti E, Amarri S, Barbato M, Barbera C, Barera G, Bellantoni A, Castellano E, Guariso G, Limongelli MG, Pellegrino S, Polloni C, Ughi C, Zuin G, Fasano A, Catassi C; SIGENP (Italian Society of Pediatric Gastroenterology, Hepatology, and Nutrition) Working Group on Weaning and CD Risk. Introduction of gluten, HLA status, and the risk of celiac disease in children. N Engl J Med. 2014 Oct 2;371(14):1295-303. doi: 10.1056/NEJMoa1400697. PMID 25271602
- [Result] Andren Aronsson C, Lee HS, Koletzko S, Uusitalo U, Yang J, Virtanen SM, Liu E, Lernmark A, Norris JM, Agardh D; TEDDY Study Group. Effects of Gluten Intake on Risk of Celiac Disease: A Case-Control Study on a Swedish Birth Cohort. Clin Gastroenterol Hepatol. 2016 Mar;14(3):403-409.e3. doi: 10.1016/j.cgh.2015.09.030. Epub 2015 Nov 25. PMID 26453955